CLINICAL TRIAL: NCT01361711
Title: A Phase 2 Trial of Alemtuzumab-Ofatumumab Combination in Previously Untreated Symptomatic Chronic Lymphocytic Leukemia
Brief Title: Alemtuzumab-Ofatumumab in Previously Untreated Symptomatic Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: GlaxoSmithKline (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Shuo Ma, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 10H06; NCI-2011-00514 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00044115 (Other: Northwestern University IRB)
Record Dates: First submitted 2011-05-16; First posted 2011-05-27 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; ofatumumab; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (monoclonal antibody therapy) (Experimental): Patients receive alemtuzumab SC three times a week in weeks 1-18 and ofatumumab IV over 4-6 hours on day 1 of weeks 3, 5, 7, 9, 11, 13, 15, and 17.
  Interventions: Biological: alemtuzumab; Biological: ofatumumab; Procedure: biopsy

INTERVENTIONS:
Biological: alemtuzumab — Given SC
  Other Names: anti-CD52 monoclonal antibody; Campath-1H; MoAb CD52; Monoclonal Antibody Campath-1H; Monoclonal Antibody CD52
Biological: ofatumumab — Given IV
  Other Names: Arzerra; HuMax-CD20
Procedure: biopsy — Correlative studies
  Other Names: biopsies

SUMMARY:
This phase II trial studies the side effects and how well giving alemtuzumab and ofatumumab together works in treating patients with previously untreated chronic lymphocytic leukemia (CLL). Monoclonal antibodies, such as alemtuzumab and ofatumumab, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer killing substances to them. Giving alemtuzumab together with ofatumumab may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the efficacy and safety of alemtuzumab-ofatumumab combination treatment in previously untreated CLL.

OUTLINE:

Patients receive alemtuzumab subcutaneously (SC) three times a week in weeks 1-18 and ofatumumab intravenously (IV) over 4-6 hours on day 1 of weeks 3, 5, 7, 9, 11, 13, 15, and 17.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have a confirmed diagnosis of CLL as defined by the International Workshop on CLL (iwCLL) 2008 (iwCLL2008) criteria below:
* Presence of at least 5x10^9 B lymphocytes/L (5000/uL) in the peripheral blood
* Morphologically, the lymphocytes must appear of small to moderate size with < 55% prolymphocytes, atypical lymphocytes or lymphoblasts
* The clonality and immunophenotype of the circulating B-lymphocytes must be confirmed by flow cytometry to express CD5, CD23, CD19, CD20, CD52 and either kappa or lambda light chain
* Patients must have symptomatic disease requiring therapy; indications for therapy are defined by the iwCLL2008 criteria as follows (one or more are sufficient):
* Clinical manifestations (if believed by the investigator to be caused by CLL): a) Unintentional weight loss > 10% within the previous 6 months; b) significant fatigue; c) fevers of greater than 100.5 degrees Fahrenheit (F) (38 degrees Celsius [C]) for 2 weeks without evidence of infection; d) night sweats without evidence of infection
* Evidence of progressive marrow failure as manifested by the development or worsening of anemia (< 11 g/dl), thrombocytopenia (< 100,000/mm^3) or neutropenia (< 1,500/mm^3)
* Massive (i.e. > 6 cm below left costal margin) or progressive splenomegaly
* Massive nodes/clusters (> 5 cm) or progressive symptomatic adenopathy
* Progressive lymphocytosis with an increase of > 50% over 2 month period, or an anticipated doubling time of less than 6 months
* NOTE: Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease is not sufficient for protocol therapy
* Patients must have evidence of adequate bone marrow reserve as shown by absolute neutrophil count (ANC) of at least 1,000/mm^3; however, if the cytopenias are due to extensive bone marrow involvement by CLL, patients may be included in the study
* And patients must have evidence of adequate bone marrow reserve as shown by platelet count of at least 50,000/mm^3; however, if the cytopenias are due to extensive bone marrow involvement by CLL, patients may be included in the study
* Serum creatinine must be less than 2.0 mg/dl obtained within 2 weeks prior to study enrollment; if serum creatinine is greater than 1.5 mg/dl, the creatinine clearance calculated from a 24 hour urine collection must be greater than 40 ml/min
* Total bilirubin must be less than 2 mg/dl (unless due to CLL involvement of liver or a known history of Gilbert's disease)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) must be no more than 2.5 times upper limit of normal unless due to disease involvement of the liver
* Alkaline phosphatase must be no more than 2.5 times upper limit of normal unless due to disease involvement of the liver
* All patients must have given a signed, informed consent prior to enrollment on study

Exclusion Criteria:

* Prior cytotoxic therapies are NOT allowed; the only exception is prior corticosteroid therapy (prednisone up to 1 mg/kg for =< 3 months) which must be stopped at least 1 week prior to study enrollment
* Patients with active autoimmune anemia or autoimmune thrombocytopenia are NOT eligible
* Patients who have current active hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver involvement by CLL, or stable chronic liver disease per investigator assessment) are NOT eligible
* Patients with active chronic or current infections requiring oral or intravenous antibiotics are NOT eligible for enrollment to the study until resolution of the infection and completion of therapeutic antibiotics
* Patients with a past or current second malignancy are NOT eligible aside from the following exceptions:
* Patients who have been free of malignancy for at least 5 years
* Patients who have a history of completely resected basal or squamous cell skin cancer, successfully treated in situ carcinoma of the breast or cervix, or pre-cancerous lesions of the colon
* Patients with known human immunodeficiency virus (HIV) are NOT eligible for the study
* Patients with history of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae are NOT eligible for the study
* Patients with clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to enrollment, congestive heart failure (New York Heart Association [NYHA ] III-IV), and arrhythmia unless controlled by therapy (with the exception of extra systoles or minor conduction abnormalities), are NOT eligible
* Patients with significant concurrent, uncontrolled medical condition including, but not limited to, cardiovascular, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient, are NOT eligible
* Patients with positive serology for Hepatitis B (HB), defined as a positive test for HB surface antigen (HBsAg), are NOT eligible; if negative for HBsAg but HB core antibody (HBcAb) positive a HB deoxyribonucleic acid (DNA) test will be performed; if HB DNA test is positive the patient is NOT eligible; NOTE: patients who are positive for HBcAb but negative for hepatitis B virus (HBV) antigenemia and viremia (HBsAg negative and HB DNA test negative) may be eligible for the study, but must be started on HBV suppression therapy with lamivudine or equivalent anti-HBV agents throughout the treatment and for a year after the completion of the treatments; these patients need to have liver function tests (LFTs) and HBV viral titer monitoring at least monthly during the treatment and for a year after treatment completion
* Patients with positive serology for hepatitis C are NOT eligible
* Women of childbearing potential and sexually active males must commit to the use of adequate contraception from the study start to one year after the last dose of study treatment
* Childbearing potential is defined as any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Adequate contraception is defined as hormonal birth control, intrauterine device, barrier method or total abstinence; patients who are unable or unwilling to use adequate contraception are NOT eligible
* Women who are pregnant or lactating are NOT eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-06; Primary Completion 2015-08-17 (Actual); Study Completion 2027-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Ma, MD, PhD, Principal Investigator — Northwestern University
Locations (2):
- Northwestern University, Chicago, Illinois, United States
- Karolinska University Hospital Solna, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened for accrual on June 3, 2011 with goal of 60 patients. First patient started treatment June 13, 2011. Accrual was suspended Sep. 26, 2011 for safety analysis of the first 6 patients. The study opened May 4, 2012 for safety cohort of 6 more patients. Study was suspended July 23, 2012 for safety analysis, and opened again Feb 4, 2013. The study closed Sep 13, 2016 because the total accrual goal for Northwestern University was met.
Groups:
- Alemtuzumab + Ofatumumab: Alemtuzumab: Administered subcutaneously, 3 times per week for up to 18 weeks at a standard dose of 30mg (except for week 1 which will dose escalate from 3mg→10mg→30mg).
  Ofatumumab: Starting at week 3, administered intravenously on day 1 of every other week prior to alemtuzumab for a total of 8 doses. For week 3 (dose 1) ofatumumab will be given at a dose of 300mg; for weeks 5, 7, 9, 11, 13, 15, and 17 (doses 2-8) ofatumumab will be given at a dose of 2000mg.
  Toxicity was assessed after completion of the extended safety run-in period of the first 12 patients at an ofatumumab dose of 2000 mg for doses 2-8. Depending on the number of patients who experienced a dose limiting toxicity in the initial 2 safety cohorts, ofatumumab doses 2-8 could have been continued at 2000 mg or reduced to 1000 mg for subsequent patients. Based on the toxicity data of the first 12 patients, ofatumumab doses 2-8 were given at 2000 mg for doses 2-8 for all patients.
  Based on experience with the initial safety run-in cohort of 6 patients, early stopping is necessary to avoid over-treatment in patients who have achieved a complete remission early. As soon as a patient is determined to have achieved MRD- CR or CRi (per iwCLL2008 criteria), both alemtuzumab and ofatumumab will be stopped.
Period: Trial Entry (Registration)
Arm/Group | Alemtuzumab + Ofatumumab
Started | 53
Received Dose of Study Drug | 52
Completed | 52
Not Completed | 1
Not completed — Patient did not meet Protocol criteria for trial entry | 1
Period: Week 9 Bone Marrow Response Assessment
Arm/Group | Alemtuzumab + Ofatumumab
Started | 52
Completed (As soon as a patient is determined to have achieved Minimal Residual Disease negative Complete Remission or Complete remission with incomplete marrow recovery (per iwCLL2008 criteria), both alemtuzumab and ofatumumab will be stopped.) | 51
Not Completed | 1
Not completed — Complete Remission in Week 8 | 1
Period: Continued Treatment After 9 Weeks
Arm/Group | Alemtuzumab + Ofatumumab
Started | 51
Completed (As soon as a patient is determined to have achieved Minimal Residual Disease negative Complete Remission or Complete remission with incomplete marrow recovery (per iwCLL2008 criteria), both alemtuzumab and ofatumumab will be stopped.) | 44
Not Completed | 7
Not completed — Complete Remission in Week 9 | 7
Period: Continued Treatment After 12 Weeks
Arm/Group | Alemtuzumab + Ofatumumab
Started (A bone marrow biopsy will be performed during week 9 to assess response. If biopsy results show residual CLL with minimal involvement (< 10% involvement), an additional bone marrow biopsy is recommended after week 12 of treatment.) | 44
Completed (As soon as a patient is determined to have achieved Minimal Residual Disease negative Complete Remission or Complete remission with incomplete marrow recovery (per iwCLL2008 criteria), both alemtuzumab and ofatumumab will be stopped.) | 41
Not Completed | 3
Not completed — Complete Remission in Week 12 | 2
Not completed — Progressive Disease at Week 11 | 1
Period: Completed Week 18 of Treatment
Arm/Group | Alemtuzumab + Ofatumumab
Started | 41
Completed (As soon as a patient is determined to have achieved Minimal Residual Disease negative Complete Remission or Complete remission with incomplete marrow recovery (per iwCLL2008 criteria), both alemtuzumab and ofatumumab will be stopped.) | 30
Not Completed | 11
Not completed — Complete Remission | 2
Not completed — Other | 9
Period: 10 Year Follow-up
Arm/Group | Alemtuzumab + Ofatumumab
Started | 52 (All patients who receive at least one dose of study drug go into follow-up.)
Completed | 2
Not Completed | 50
Not completed — Still in follow-up | 22
Not completed — Death | 7
Not completed — Developed new cancer | 1
Not completed — Lost to Follow-up | 2
Not completed — New treatment started | 6
Not completed — Progressive Disease and New treatment started | 11
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Groups:
- Alemtuzumab + Ofatumumab: Alemtuzumab: Administered subcutaneously, 3 times per week for up to 18 weeks at a standard dose of 30mg (except for week 1 which will dose escalate from 3mg→10mg→30mg).
  Ofatumumab: Starting at week 3, administered intravenously on day 1 of every other week prior to alemtuzumab for a total of 8 doses. For week 3 (dose 1) ofatumumab will be given at a dose of 300mg; for weeks 5, 7, 9, 11, 13, 15, and 17 (doses 2-8) ofatumumab will be given at a dose of 2000mg.
  Toxicity was assessed after completion of the extended safety run-in period of the first 12 patients at an ofatumumab dose of 2000 mg for doses 2-8. Depending on the number of patients who experienced a dose limiting toxicity in the initial 2 safety cohorts, ofatumumab doses 2-8 could have been continued at 2000 mg or reduced to 1000 mg for subsequent patients. Based on the toxicity data of the first 12 patients, ofatumumab doses 2-8 were given at 2000 mg for doses 2-8 for all patients.
  biopsy: Correlative studies
Arm/Group | Alemtuzumab + Ofatumumab
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 20
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Best Response as Defined by the iwCLL2008 (International Workshop on Chronic Lymphocytic Leukemia 2008)
Description: CR= Absence of clonal lymphocytes in the peripheral blood, significant lymphadenopathy, hepatomegaly or splenomegaly, and constitutional symptoms. Blood counts: Neutrophils ≥ 1,500/μL; Platelets >100,000μL; Hemoglobin > 11.0g/dL. Bone marrow normocellular for age, less than 30% of nucleated cells = lymphocytes. Lymphoid nodules absent. CRi= Fulfills CR but anemia or thrombocytopenia or neutropenia related to drug toxicity. PR= 2 criteria from group A and 1 from Group B. Group A: Decrease in the number of blood lymphocytes of 50% or more. Reduction in lymphadenopathy. No increase in any lymph node, and no new enlarged lymph node. A decrease in liver by at least 50% from baseline. Decrease in the size of the spleen by 50% or more. Reduction in marrow infiltrate or B-lymphoid nodules. Group B: Platelet counts > than 100,000/μL or 50% better. Hemoglobin > than 11.0g/dL or 50% better. Neutrophils>1500/μL or 50% better. Criteria is continued in Analysis Population Description below...
Time Frame: Range of responses between 8 weeks from initiation of treatment to 2 months post-treatment.
Population: Criteria from Outcome Measure Description cont. MRD=Bone marrow with less than one CLL cell per 10,000 leukocytes. To qualify as a PD: at least two of the criteria of in Group A, plus one of the criteria in Group B, must be met. Group A: An increase ≥ 50% of: lymphadenopathy, hepatomegaly, or splenomegaly. An increase ≥ 50% over baseline in blood lymphocytes. Group B: Platelet count decrease of ≥ 50% from baseline secondary to CLL, Hemoglobin decrease of > 2g/dl from baseline secondary to CLL.
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab + Ofatumumab
Number analyzed (Participants) | 52
Participants
  Complete Remission (CR), Minimal Residual Disease (MRD) Negative | 18
  Complete Remission (CR), Minimal Residual Disease (MRD) positive | 2
  Complete Remission, MRD status unknown | 3
  Complete Remission with Incomplete Marrow Recovery (CRi) | 2
  Partial Remission (PR) | 26
  Progressive Disease (PD) | 1

2. Secondary Outcome: Survival Rates
Description: Survival rates will be calculated for progression-free survival (PFS), therapy-free survival (TFS), and overall survival (OS).
Time Frame: Up to 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Treatment Toxicity as Measured by Adverse Events Experienced While on Treatment
Time Frame: Weeks 1, 3, 5, 7, 9, 11, 13, 15, and 17
Reporting Status: Not Posted

4. Secondary Outcome: Correlation of Disease Characteristics With Disease Outcomes
Description: Clinical outcomes (such as response, PFS and TFS) will be correlated with pre-treatment clinical and biological characteristics(such as Rai staging, presence of bulky lymph nodes, cytogenetics by FISH, CD38, ZAP70 and IgVH mutation status).
Time Frame: At baseline and over 18 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Compare Efficacy Between This Study and Historical Control Study of Alemtuzumab-rituximab
Description: Response and survival rates will be compared between the two studies.
Time Frame: At baseline and over 18 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a four year period. Each patient was followed from the time of treatment, and during treatment up to 18 weeks. Adverse events were collected up to 60 days post-therapy. Serious adverse events (SAEs) were collected for one year after treatment discontinuation or until the initiation of second-line therapy.
Arm/Group | Alemtuzumab + Ofatumumab
All-Cause Mortality (participants affected / at risk) | 6/52
Serious Adverse Events (participants affected / at risk) | 20/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab + Ofatumumab (N=52)
Infection (Infections and infestations) | 1
Abnormal Platelets (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 4
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Fever (General disorders) | 3
CMV infection (Infections and infestations) | 1
MRSA Bacteremia (Infections and infestations) | 1
Neutropenic fever (Blood and lymphatic system disorders) | 1
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1 — This patient also experienced hypercalcemia at the time of this event.
Sinus tachycardia (Cardiac disorders) | 1
Meningitis (Infections and infestations) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Allergic reaction (Immune system disorders) | 1 — The patient also experienced fever at the time of this event.
CMV positive (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Lung infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab + Ofatumumab (N=52)
Abdominal cramping (Gastrointestinal disorders) | 1
Abdominal discomfort (General disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abnormal C-reactive protein levels (Investigations) | 1
Abnormal Hemoglobin count (Investigations) | 44
Abnormal neutrophil count (Investigations) | 44
Abnormal platelet count (Investigations) | 43
Abscess (Infections and infestations) | 1
Actinic keratoses (Skin and subcutaneous tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase increased (Investigations) | 14
Alkaline phosphatase increased (Investigations) | 8
Allergic reaction (Immune system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 3
Appendicitis (Infections and infestations) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 24
Atrial fibrillation (Cardiac disorders) | 1
Autoimmune disorder (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Basal Cell Carcinoma Recurrence (Investigations) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Blood bilirubin increased (Investigations) | 3
Blurred vision (Eye disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Borderline diabetes (Metabolism and nutrition disorders) | 1
Brown tint to vision (Eye disorders) | 1
Cerumen Impaction (Ear and labyrinth disorders) | 1
Cherry angiomas (Skin and subcutaneous tissue disorders) | 1
Chest pain (Cardiac disorders) | 1
Chest tightness (General disorders) | 2
Chills (General disorders) | 13
High cholesterol (Investigations) | 1
CMV reactivation (Infections and infestations) | 18
CMV Infection (Infections and infestations) | 11
Concentration impairment (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Coronary artery disease (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine increased (Investigations) | 16
Cytokine release syndrome (Immune system disorders) | 2
Decrease absolute CD3+ (Investigations) | 1
Decrease absolute CD3+CD8+ (Investigations) | 1
Decrease absolute CD3+CD4+ (Investigations) | 1
decreased hematocrit (Investigations) | 1
Decreased B cell % (Investigations) | 1
Decreased IgG (Blood and lymphatic system disorders) | 1
Decreased IgA (Blood and lymphatic system disorders) | 1
Decreased IgM (Blood and lymphatic system disorders) | 1
Decreased urination (Renal and urinary disorders) | 1
Depression (Psychiatric disorders) | 2
Diabetes (Metabolism and nutrition disorders) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 15
Diffuse Large B-Cell Lymphoma (Blood and lymphatic system disorders) | 1
Diverticulosis (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 4
Double vision (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Easy bruising (Blood and lymphatic system disorders) | 1
Edema limbs (General disorders) | 4
Elevated LDH (Investigations) | 7
Elevated neutrophils (Blood and lymphatic system disorders) | 1
Elevated Quantitative IgG (Immune system disorders) | 1
Enlarged adrenal glands (Endocrine disorders) | 1
Enlarged lymph node in left groin (Investigations) | 1
Enlargement of prostate gland (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Erythematous Rash (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 34
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Fever (General disorders) | 35
Flu like symptoms (General disorders) | 12
Flushing (Vascular disorders) | 1
Gait disturbance (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Genital herpes (Infections and infestations) | 1
guttate psoriasis (Skin and subcutaneous tissue disorders) | 1
Headache (General disorders) | 2
Headache (Nervous system disorders) | 4
Hemolysis (Blood and lymphatic system disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hepatitis B positive (Hepatobiliary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 25
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hyperlipidemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 9
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypogammaglobulinemia (Immune system disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyposmia (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
IgM paraprotein (Investigations) | 1
Increased C-reactive protein. (Investigations) | 1
Infusion related reaction (General disorders) | 29
Infusion site extravasation (General disorders) | 2
Injection site reaction (General disorders) | 47
Insomnia (Psychiatric disorders) | 2
Iron deficiency (Investigations) | 1
Itchiness in throat (General disorders) | 1
Keratitis (Eye disorders) | 1
lack of vitamin B12 (Metabolism and nutrition disorders) | 1
Laparoscopic appendectomy (Surgical and medical procedures) | 1
Left branch bundle block (Cardiac disorders) | 1
Left lumbar spasm (Musculoskeletal and connective tissue disorders) | 1
Legionella Pneumonia (Infections and infestations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lightheadedness (General disorders) | 1
Lower leg lesions (Skin and subcutaneous tissue disorders) | 1
Lung infection (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 24
Lymphocyte count increased (Investigations) | 3
Malaise (General disorders) | 2
Memory impairment (Nervous system disorders) | 1
Meningitis (Infections and infestations) | 1
MRSA Bacteremia (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 9
Neutrophil count decreased (Investigations) | 3
Night Sweats (General disorders) | 11
Nonspecific T Wave Abnormalities (Cardiac disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pain in shoulder (Musculoskeletal and connective tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palpitations (Cardiac disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral neuropathy in feet (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8
perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1
Petechiae on upper abdomen (Skin and subcutaneous tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
pneumonia, community acquired (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pressure with urination (Renal and urinary disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Proteinuria (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pulmonary emboli (Vascular disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
redness of the skin with scaling (Skin and subcutaneous tissue disorders) | 1
Benign prostatic hyperplasia (Renal and urinary disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Ringing in ears (Investigations) | 1
Rising PSA (Investigations) | 1
Scalp psoriasis (Skin and subcutaneous tissue disorders) | 1
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1
Seborrheic keratoses (Skin and subcutaneous tissue disorders) | 1
Sensory numbness (Nervous system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Skin tear on right buttock (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Spongiotic Dermatitis (Skin and subcutaneous tissue disorders) | 1
Subacute Spongiotic Dermatitis (Skin and subcutaneous tissue disorders) | 1
Sun damaged skin (Skin and subcutaneous tissue disorders) | 1
Surgery for testicular varicose (Surgical and medical procedures) | 1
surgery to remove two small basiliom (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Thromboembolic event (Vascular disorders) | 5
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Tinea pedis (Skin and subcutaneous tissue disorders) | 1
Tingling in fingertips to elbows (Nervous system disorders) | 1
Tingling in lips (Nervous system disorders) | 2
Tingling in the face (Skin and subcutaneous tissue disorders) | 1
Tonsillectomy (Surgical and medical procedures) | 2
Upper respiratory infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 1
Vaginal Atrophy (Reproductive system and breast disorders) | 1
Vaginal infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 35
Worsening of gout (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The participating site (Karolinska University Hospital Solna) did not meet the total accrual goal. However, the lead site (Northwestern University) did.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes